CLINICAL TRIAL: NCT03343275
Title: Multicenter, Controlled and Randomized Clinical Trial to Evaluate the Combined Use of a Medical Device and a Food Supplement in the Control of Urinary pH in Patients With an Implanted Double Pigtail Stent
Brief Title: Combined Use of a Medical Device and a Dietary Complement in Patient Urinary pH Control in Patients With an Implanted Double J Stent.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Devicare S.L. (Industry)
Collaborators: Clever Instruments S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DEV-LCD-02-17
Record Dates: First submitted 2017-11-02; First posted 2017-11-17 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Stent Complications
Keywords: Stent, incrustation, pH Control

STUDY DESIGN:
Intervention Model Description: Adults attending urology/nephrology consultation whom have been recently implanted a double J stent or have its implantation programmed and are able of taking care in urinary pH self-control.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Dietary supplement : Lit-Control® pH Down
  * Pharmaceutical form: capsules
  * Administration : oral
  * Dose: 3 capsules/day.
    • Sanitary product : Lit-Control® pH Meter
  * In vitro diagnosis sanitary product
  * Use:Urinary pH evaluation
  Interventions: Combination Product: Lit control pHDown
- Placebo (Placebo Comparator): Placebo:
  * Pharmaceutical form: capsules
  * Administration : oral
  * Dose: 3 capsules/day.
    • Sanitary product : Lit-Control® pH Meter
  * In vitro diagnosis sanitary product
  * Use:Urinary pH evaluation
  Interventions: Combination Product: Lit control pHDown

INTERVENTIONS:
Combination Product: Lit control pHDown — Patients within the experimental arm will receive dietary supplement Lit-control®pH Down to help them keep their urinary pH in the adequate levels, being these considered as the preventive ones to avoid stent calcification (pH<6.2) being the 3 capsule per day indication. On the other hand, the control arm will receive a placebo product with similar organoleptic qualities and the same posology characteristics. Both arms wil use Lit-Control® pH Meter device to keep self- control of the urinary pH; also, both will receive the same hygienic-dietary indications about the care of the stent.

SUMMARY:
This study evaluates the effectivity in urinary pH Control and the prevention of calcification in Double J stent using a device combined with the intake of dietary supplements. Every patient will receive hygienic-dietary indications.

Patients will also take one out of the three dietary supplements regarded within the study (pH Up, pH Down and Cysteine) to control the adequate pH level, always following medical indications.

DETAILED DESCRIPTION:
Several studies have shown the importance of urinary pH Control (pHv) to determine the frequency of stent incrustation, this measure being a variable to be taken into account in the management of catheterized patients. However, the level of pHv is influenced by multiple factors, so its routine control is difficult to interpret. The nucleation pH (pHn) was described on 1999: the pH where the incrustation starts to form. In his study he observed that the pH of the patients who developed a stent blockage and the pH of those who were not very similar (7.46 and 7.38 respectively), but observed that the pHv of the patients who did not have incrustations was much lower and therefore had a much wider safety margin.

As already mentioned, pHv is influenced by different factors, but it is especially sensitive to diet. For this reason, hygienic and dietetic interventions (exercise, diet, fluid intake, etc.) are one of the preventive measures of incrustation of the stent of great utility, although its effectiveness is subject to patient adherence.

Lit-control®pH Down is a dietary supplement with an acidifying effect on urine, which helps in the prevention of complications arising from the alkalinization of urine. It contains L-methionine, phytin (calcium-magnesium phytate salt), zinc and vitamin A. The two active components in pHv acidification are L-methionine and phytin,while zinc and vitamin A increase the action of phytin. Specifically, zinc favors the affinity of its affinity for calcium phosphate and vitamin A prevents its degradation by alkaline phosphatase.

L-methionine is an essential amino acid that plays an important role in metabolic processes. It is normally acquired through food and absorbed in the small intestine to be metabolized in the liver via cysteine to sulphate and protons. Consequently, its administration produces a significant reduction of urinary pH.

According to the European Association of Urology (UAE), urinary acidification with L-methionine up to pH 5.8 - 6.2 is recommended as a therapeutic measure for calculations of struvite, calcium phosphate and ammonium urate at doses of 600- 1500 mg / day. This recommendation is based on the results observed in 1996, where an acidification of the pH of the urine of the patients was observed from 7.5 to 5.5 after the administration of 1500-3000 mg / day (3-6 capsules) of 500mg / day. Also in the study of Hesse 1999 a significant reduction in urinary pH was observed up to pH = 6.0 after the administration of a single dose of 1500 mg of L-methionine, maintaining this effect for 24h. In addition, a significant reduction was observed versus the control group in terms of the relative supersaturation for struvite and brushite in the urine of 24h. In another more recent study, the authors studied the circadian course of urinary pH after the administration of 1500 mg of L-methionine. They observed a strong decrease in urinary pH up to 2h after the administration of the amino acid that remained at significantly low levels for 8h, resulting in a pH level for 24h between 5.98 and 6.32. Therefore, in order to guarantee therapeutic doses of L-Methionine (1500mg / day), the Lit-control®pH Down regimen to follow would be equivalent to 3 capsules per day (500 mg / capsule).

On the other hand, the device Lit-control® pH Meter is a medical device that allows patients to self-monitor their pHv daily in their own home, allowing a thorough control of the pH and the level of risk of incrustation. The device has been validated for use in lithiasic patients, with applicability in the treatment of other urological pathologies related to the acid-base balance of urine, calcifications of urinary stents, cystitis, urinary tract infections, painful bladder syndrome and bladder hyperactive

The objective of this study is to evaluate the effectiveness of the food supplement Lit-control®pH Down in the prevention of double J stent incrustation and in the control of urinary pH together with the use of the device Lit-control® pH meter

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patients which have been recently implanted a Double J stent (less than a week implant) or who have planned their implant and have been recommended with pH control to avoid incrustation/calcification.
* Patients who accept their participation in the study and give their informed consent

Exclusion Criteria:

* Patients with base pathologies wich , based on clinical criteria, aren´t sensitive about the study dietary supplement indications.
* Patients which have programmed the stent extraction 3 weeks before base visit.
* Uric and cystinuric patients which requires pH control different from the established study protocol .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Incrustation Score | 2 days
  0 (No incrustation); 1(Sporadic incrustation less than 1-2 mm); 2 (Wide area calcifications more than 1-2 mm) ; 3 (Total obstruction)
Urinary pH level | 2 times/day
Stent implant cause | 2 months
  Medical evaluation and diagnosis leading to stent implant
Self-control below values 6.2 | 2 times/day

SECONDARY OUTCOMES:
Anatomic alterations on the urinary system | 2 months
  Medical evaluation on the different alterations present in the urinary system.
Previous uropathic obstructive incidence | 2 months
  Number of obstructions in the past two months.
Date of past stent implants | 2 months
pH control: Total time | 2 times/day
2 hours urine analysis :Fasting | 2 hours
Urine culture | 48 hours
Complications associated with stent implant | 2 months
Treatment adherence | 2 months
  The clinical will evaluate the patient treatment adherence by means of Morisky-Green test
Stent extraction data | 2 months
  Possibility of complications during the extraction, date of extraction, intervention type, intervention duration
Blockage risk factor | 1 month prior intervention
  Evaluation by clinical evaluation
Date of stent extraction | 2 months
Type of previous stent | 2 months
  Description of the previous stent
Number of different symptoms associated with the previous calcification | 2 months
  Different symptomatology associated with the previous calcification

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Universitario de Valme, Seville, Andalusia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Fundació Puigvert, Barcelona
  - Hospital Clínico Universitario San Cecilio, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Rio Hortega, Valladolid

REFERENCES:
- [Derived] Torrecilla C, Fernandez-Concha J, Cansino JR, Mainez JA, Amon JH, Costas S, Angerri O, Emiliani E, Arrabal Martin MA, Arrabal Polo MA, Garcia A, Reina MC, Sanchez JF, Budia A, Perez-Fentes D, Grases F, Costa-Bauza A, Cune J. Reduction of ureteral stent encrustation by modulating the urine pH and inhibiting the crystal film with a new oral composition: a multicenter, placebo controlled, double blind, randomized clinical trial. BMC Urol. 2020 Jun 5;20(1):65. doi: 10.1186/s12894-020-00633-2. PMID 32503502

DOCUMENTS (1):
  • Study Protocol (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT03343275/Prot_001.pdf